CLINICAL TRIAL: NCT02246933
Title: Effects of a PUFA-rich Diet on Acute Metabolic and Inflammatory High-Fat Meal Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Jamie Cooper, Associate Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 503815
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Inflammation; Obesity
MeSH Terms: conditions — Inflammation; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PUFA Diet (Experimental)
  Interventions: Other: PUFA Diet
- Control Diet (Placebo Comparator)
  Interventions: Other: Control Diet

INTERVENTIONS:
Other: PUFA Diet — The 7-day diet will consist of 50% carbohydrate, 15% protein, and 35% fat. 21% of total energy will be poly-unsaturated fatty acids, 9% mono-unsaturated fatty acids, and 5% saturated fatty acids.
  Arms: PUFA Diet
Other: Control Diet — The 7-day diet will consist of 50% carbohydrate, 35% fat, and 15% protein. Furthermore, 7% of total energy will be poly-unsaturated fatty acids, 15% of total energy will be mono-unsaturated fatty acids, and 13% of total energy will be saturated fatty acids.
  Arms: Control Diet

SUMMARY:
This study evaluates whether a diet rich in poly-unsaturated fats can compensate for the negative effects of high saturated fat meals on metabolic, inflammatory, and coagulation responses. Half of the participants will receive a high polyunsaturated fat diet )50% carbohydrate, 15% protein, and 35% fat. 21% of total energy will be poly-unsaturated fatty acids, 9% mono-unsaturated fatty acids, and 5% saturated fatty acids) for 7 days, while the other half will receive a control diet 50% carbohydrate, 35% fat, and 15% protein 50% carbohydrate, 35% fat, and 15% protein. Only, 7% of total energy will be poly-unsaturated fatty acids, 15% of total energy will be mono-unsaturated fatty acids, and 13% of total energy will be saturated fatty acids.) for 7 days.

DETAILED DESCRIPTION:
Eating more saturated fats has been shown to decrease how many calories an individual burns and increase chronic disease risk by increasing inflammation, coagulation (blood clotting) potential, blood pressure, and cholesterol. Conversely, eating more poly-unsaturated fats has been linked to decreased risk of chronic diseases. The goal of this study is to determine whether or not eating a diet containing a lot of poly-unsaturated fats can compensate for the damaging effects of eating occasional high-fat meals that are high in saturated fats. Those damaging effects we are interested in studying include how much fat and calories a person's body burns, and measuring some markers of chronic disease risk in the blood (inflammation markers and blood clotting markers).

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women between the ages of 18 and 45y with a normal weight based on body mass index (BMI=18-24.9kg/m2), must be sedentary (perform less than 3 hours per week of structured exercise) and , if participant has fasting total cholesterol >200 gm/dL, high-density lipoprotein <40 mg/dL, low-density lipoprotein cholesterol >100 mg/dL, and/or triglycerides >150 mg/dL (based on fasting blood lipids).

Exclusion Criteria:

* Weight loss or gain exceeding 5% of body weight in the past 3 months
* Current participation in a weight loss program
* Any current exercisers (greater than 3h per week)
* Any person who is on a medically prescribed diet
* Any person who is vegan, or any type of vegetarian other than pesco-vegetarian
* Any chronic or metabolic disease, hyperlipidemia, gastrointestinal disorder, or history of medical or surgical events that could affect digestion and absorption of nutrients
* Any current supplement use other than a daily multivitamin (this includes fish oil supplements)
* Any current medication use other than birth control (this includes anti-inflammatory NSAID use).
* Anyone who is pregnant, lactating, or planning a pregnancy
* Anyone who has donated blood or plasma in the last 20 days
* Any tobacco users
* Anyone who has allergies to the most common food allergens (milk, eggs, peanuts, almonds, cashews, walnuts, fish, shellfish, soy and wheat) or to any of the food that will provided during the study
* Anyone who has allergies to any of the components of the liquid meals

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Blood Markers | Change measures baseline and 9 days
  Change in inflammation and coagulation factors

SECONDARY OUTCOMES:
Change in Energy Expenditure | Change measures baseline and 9 days
Change in Substrate Oxidation | Change measures baseline and 9 days
Change in Fasting Blood Lipids | Change measures baseline and 9 days
Change in Systolic Blood Pressure | Change measures baseline and 9 days

CONTACTS AND LOCATIONS:
Overall Officials: jamie A Cooper, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia - Department of Foods and Nutrition, Athens, Georgia, United States

REFERENCES:
- [Derived] Kaviani S, Taylor CM, Stevenson JL, Cooper JA, Paton CM. A 7-day high-PUFA diet reduces angiopoietin-like protein 3 and 8 responses and postprandial triglyceride levels in healthy females but not males: a randomized control trial. BMC Nutr. 2019 Jan 6;5:1. doi: 10.1186/s40795-018-0262-7. eCollection 2019. PMID 32153916